CLINICAL TRIAL: NCT01065727
Title: Study Impact, on Clinical Outcomes, Quality of Life and Costs of 2 Therapeutic Strategy (Monthly Natalizumab Versus Mitoxantrone Then Immunomodulator) at 3 Years of Follow-up for Aggressive Remitting Multiple Sclerosis
Brief Title: Impact Study of 2 Therapeutic Strategy for Aggressive Remitting Multiple Sclerosis
Acronym: IQUALYSEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PHRC/09-06
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Multiple Sclerosis
Keywords: Reemitting aggressive multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mitoxantrone followed by immunomodulator (Experimental)
  Interventions: Other: mitoxantrone - immunomodulator
- natalizumab (Active Comparator)
  Interventions: Other: natalizumab

INTERVENTIONS:
Other: mitoxantrone - immunomodulator — mitoxantrone during 6 months and followed by immunomodulator during 2 years and half
  Arms: mitoxantrone followed by immunomodulator
Other: natalizumab — monthly natalizumab during 3 years
  Arms: natalizumab

SUMMARY:
Cost-effectiveness study of 2 disease-modifying therapies (natalizumab versus mitoxantrone followed by immunomodulator) in the management of aggressive remitting multiple sclerosis

ELIGIBILITY:
Inclusion Criteria:

* Patients with remitting multiple sclerosis according to mac Donald criteria
* aggressive remitting multiple sclerosis according to following criteria:
* 2 or less disabling relapse during the 12 months before inclusion
* 1 or more
* EDSS between 2 and 5
* aged less or equal to 40 years old for the women
* effective contraception

Exclusion Criteria:

* patients less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2010-02; Primary Completion 2016-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
cost effectiveness | 30 years

SECONDARY OUTCOMES:
progressive neurological disability | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Edan Gilles, MD PhD, Principal Investigator — Rennes University Hospital
Locations (2):
- France (2):
  - CHU Cavale Blanche, Brest
  - CHU Rennes, Rennes